CLINICAL TRIAL: NCT04140019
Title: Early Cardiac Magnetic Resonance Imaging in Suspected Non-ST-Elevation Myocardial Infarction: An Observational Two-Center Study
Brief Title: Early Cardiac Magnetic Resonance Imaging in Suspected Non-ST-Elevation Myocardial Infarction
Acronym: CMR-OBSERVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: NL65125.068.18
Record Dates: First submitted 2019-08-13; First posted 2019-10-25 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: NSTEMI - Non-ST Segment Elevation MI; ACS - Acute Coronary Syndrome
Keywords: NSTEMI; NSTE-ACS; CMR; Troponin T; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSTEMI
  Interventions: Diagnostic Test: CMR

INTERVENTIONS:
Diagnostic Test: CMR — Early CMR with adenosine stress/rest perfusion before invasive coronary angiography.

SUMMARY:
Background and rationale: Evaluating patients with acute chest pain, elevated high-sensitive cardiac troponin (hs-cTn) levels and non-diagnostic electrocardiogram (ECG), i.e. suspected non-ST elevation myocardial infarction (MI), is a daily challenge. Although contemporary hs-cTn assay-based algorithms have greatly facilitated clinical decision-making, still one-quarter of patients is categorized as 'observe' group and in whom a diagnosis initially remains unknown. Although routinely treated as acute (MI) with referral to invasive coronary angiography (ICA), up to one-third does not have obstructive coronary artery disease (CAD). Follow-up cardiac magnetic resonance imaging (CMR) has been shown to be a very useful diagnostic tool in this setting but is not part of routine clinical care in every patient.

Objectives: To investigate in patients with suspected non-ST elevation MI meeting the 'observe' criteria and who are scheduled for ICA: 1) the prevalence of coronary artery disease as well as non-coronary artery disease related and extra-cardiac diseases by adding CMR early in the diagnostic pathway, and 2) the number of major adverse cardiac events (MACE) and a composite of MACE and major (non-cardiac) adverse events after 30 days and one year. These objectives allow an accurate estimate of the number of potentially avoidable ICA in the future and whether early CMR could be a safe gatekeeper for inappropriate ICA.

Study population and design: In this prospective, observational two-center study in The Netherlands (MUMC+ and VieCuri Medical Center), 87 consecutive patients with acute chest pain, non-diagnostic ECG and hs-cTn levels meeting the observe criteria and scheduled for ICA, will be investigated. Patients will undergo a comprehensive CMR examination prior to ICA and will be followed-up at one month and one year. After completion of follow-up, an independent clinical diagnosis committee will adjudicate a final diagnosis: at discharge and after one year. The final diagnosis at discharge will be adjudicated twice: once with and once without considering the results of CMR. For the diagnosis at one-year, all clinical variables and CMR results will be considered. MACE and complications will be scored after 30 days and one year.

Main study parameters/endpoints: The primary endpoint is the prevalence of coronary artery disease as well as non-coronary artery disease related and extra-cardiac diseases. The secondary (safety) endpoint is the number of major adverse cardiac events (MACE) and a composite of MACE and major (non-cardiac) adverse events after 30 days and one year.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

CMR is an accepted and safe imaging modality in patients with (suspected) non-ST-elevation myocardial infarction.

DETAILED DESCRIPTION:
1. OBJECTIVES 1.1 Primary Objective To investigate the prevalence of coronary artery disease as well as non-coronary artery disease related and extra-cardiac diseases in patients presenting with acute chest pain, a non-diagnostic ECG and elevated hs-cTn levels meeting the 'observe' criteria by using CMR early in the diagnostic pathway and at least prior to intended invasive coronary angiography.

   1.2 Secondary Objective

   To investigate in patients presenting with acute chest pain, a non-diagnostic ECG and elevated hs-cTn levels meeting the 'observe' criteria and who are scheduled for ICA:
   * The number of MACE and a composite of MACE and major (non-cardiac) adverse events after 30 days and one year.
   * The diagnostic accuracy of CMR for the diagnosis of obstructive CAD (i.e. stenosis ≥70%)
2. STUDY DESIGN This prospective, two-center observational study will be performed in Maastricht University Medical Center (MUMC+) and VieCuri Medical Center, Venlo, The Netherlands. Patients visiting the cardiac ED with acute chest pain, a non-diagnostic ECG and hs-cTn levels meeting the 'observe' criteria and who are scheduled for ICA are eligible. After written informed consent, patients will be included. They will be treated according to current guidelines and undergo a comprehensive CMR investigation as soon as possible after inclusion but at least prior to an intended ICA (taking into account the guideline requirement of performing ICA <72 hours after admission). Early CMR will not interfere with routine clinical care and was previously shown to be feasible.(16) The interventional cardiologists and treating physicians will be blinded for the CMR results since this is not part of current clinical practice. All CMR studies will be analyzed in MUMC+ (i.e. core lab) as soon as possible after ICA is performed. Only incidental extra-cardiac findings that may significantly change clinical management will be reported to the treating physician (i.e. malignancy, massive pulmonary embolism, acute aortic dissection, etc.). Also, when a clinical diagnosis remains unknown after ICA and only if clinicians explicitly request to perform additional CMR as a clinical routine, the results of the early CMR will be provided. Patients will be followed at least after 30 days and one-year and normal clinical variables, final diagnosis, total number of ICA and outcome (MACE and major (non-cardiac) adverse events) will be collected in each patient. After all patients have completed their one-year follow-up, an independent final diagnosis committee will adjudicate a final diagnosis. This committee will adjudicate a final diagnosis: 1) after the index discharge, and 2) after one year. The final diagnosis at discharge will be adjudicated twice by the committee: once with and once without considering the results of CMR. For the adjudicated final diagnosis at one-year, all clinical variables including the results of CMR will be considered.

3 STUDY POPULATION

3.1 Population Patients presenting to the cardiac ED with acute chest pain, a non-diagnostic ERCG, elevated hs-cTn levels meeting the 'observe' criteria and who are admitted and scheduled for an ICA, will be eligible to participate in this study.

In MUMC+, approximately 4000 patients visit the cardiac ED every year of whom half present with acute chest pain.(25) After excluding 15% of patients with ST-Elevation Myocardial Infarction (STEMI), 1700 patients with acute chest pain need further evaluation. Approximately one-quarter (n=425) meet the 'observe' criteria.(8) Although a rather conservative estimate, based on pilot data and previous study results (25), the investigators expect that at least 20% of patients (n=90) will be eligible or willing to participate in a similar research trial per center. Because the number of cardiac ED visits in VieCuri Medical Center is comparable to MUMC+, it is expected that all 87 patients can be included within one year after start of the study.

The study will be performed according to Good Clinical Practice (GCP) guidelines and the data will be analyzed and reported in accordance with the CONSORT (Consolidated Standard of Reporting Trials) guidelines. Prior to inclusion, patients will be asked to give written informed consent.

3.2 Inclusion criteria

* Acute onset (>1 hour) chest pain (or angina pectoris equivalent) suspected of non-ST-elevation myocardial infarction (NSTEMI)
* Hospital admission and scheduling for ICA
* Hs-cTn levels meeting the 'observe' criteria
* Age between 18 years - 85 years old
* Written informed consent 3.3 Exclusion criteria
* Refractory angina or on-going severe ischemia requiring immediate ICA
* Patients requiring ICA < 24 hours after admission (see previous bullet)
* Hemodynamic instability and/or cardiogenic shock (mean arterial pressure <60 mmHg)
* Heart failure (Killip Class ≥ III) requiring intravenously medication (nitroglycerine, diuretics, etc.)
* ST-Elevation Myocardial Infarction (ST-elevation in 2 contiguous leads: ≥0.2mV in men or ≥0.15 mV in women in leads V2-V3 and/or ≥0.1 mV in other leads or new left bundle branch block)
* Symptoms highly suggestive of non-cardiac origin at presentation (as judged by the cardiac ED physician/cardiologist)
* Symptoms highly suggestive of AAD, PE, or acute peri-myocarditis
* Inability to organize ICA and CMR <72 hours after admission (especially for patients admitted on Friday evenings/nights (logistic restrictions).
* Life threatening arrhythmias prior to or during presentation (sustained ventricular tachycardia, repetitive non-sustained ventricular tachycardia, ventricular fibrillation, sinoatrial or atrio-ventricular block)
* Atrial fibrillation with persistent ventricular rate ≥100 beats per minute (bpm) after treatment
* Ongoing tachycardia (≥100/bpm)
* Angina pectoris secondary to anemia (<5.6 mmol/L), untreated hyperthyroidism, or severe hypertension (>200/110 mmHg)
* More than mild aortic and mitral valve calcification or stenosis by latest echocardiography
* Recent revascularization or ACUTE MI (<6 months)
* Known CAD not suitable for further interventions (PCI or CABG)
* Pregnancy
* Breast feeding women
* Life expectancy <1 year (malignancy, etc.)
* Refusal of data storage until 15 years after end of study
* Participation in another investigational study that has not reached its primary endpoint
* Contraindications to CMR:

ODIN-protocol: "Uitvoering van MRI-onderzoek bij patiënten met een cardiaal implanteerbaar elektronisch device (CIED), waaronder een pacemaker en ICD"; ODIN-protocol: "Voorbereiding klinische patiënten voor MRI-onderzoek"

* Metallic implant (vascular clip, neuro-stimulator, cochlear implant)
* Pacemaker or implantable cardiac defibrillator (ICD)
* Claustrophobia
* Body weight >130 kg or body habitus that does not fit into the gantry
* Renal failure (estimated Glomerular Filtration Rate (eGFR) ≤30 mL/min/1,73m2) / chronic renal failure stage 4-5
* Known severe allergy to gadolinium contrast agents (patient with mild allergy is eligible for inclusion when pre-medication according to hospital guidelines can be administered)

  • Contraindications to adenosine:
* High degree atrio-ventricular block (2nd or 3rd degree)
* Severe bronchial asthma
* Chronic obstructive pulmonary disease GOLD >=III
* Concomitant use of Dipyridamole (Persantin)
* Long QT syndrome (congenital)

3.4 Patient inclusion process Eligible patients need to have acute chest pain (or angina pectoris equivalent) for at least one hour, a non-diagnostic ECG and hs-cTn levels meeting the 'observe' criteria and need to be admitted and scheduled for ICA. The physician working on the cardiac ED will screen patients. When eligible, patients will be informed about the study and asked for oral permission to be approached by a member of the research team. Two hours after written information is given, the patient is asked to participate. After written informed consent, the patient is included in the study.

3.5 Sample size calculation This is an observational study primarily aiming to investigate the prevalence of non-coronary artery and extra-cardiac diseases in patients presenting with acute chest pain, non-diagnostic ECG and elevated hs-cTn levels meeting the 'observe' criteria (i.e. patients with suspected NSTEMI) and who are scheduled for ICA. Knowing this prevalence will help to determine the number of potentially avoidable ICA in the future.

Based on studies performed in comparable but not similar patients in the conventional troponin assay (non-hs-cTn) era, the investigators transpose a prevalence of at least 20% having non-obstructive CAD to the current population. This is a rather conservative estimation and the prevalence is expected to be even higher in the current high-sensitive troponin assay era. Similarly, the investigators transpose the results of additional CMR in patients with ST-elevation myocardial infarction and non-obstructive CAD where CMR was helpful providing a diagnosis in 70%. Using follow-up CMR in this setting, myocarditis can be diagnosed in 34%, (stress) cardiomyopathy in 15%, PE or AAD in 1%, and other diseases in 2% of patients. Interestingly, MI or myocardial ischemia can still be diagnosed in 20% of patients in the absence of obstructive CAD. CMR is expected to be normal in 25% and non-diagnostic in 5%.

ICA will be considered appropriate when obstructive CAD is found at ICA and, for safety reasons, when CMR shows MI or myocardial ischemia despite non-obstructive CAD at follow-up ICA (in 20%) or when CMR is non-diagnostic (in 5%). The total proportion of appropriate ICA is thus expected to be 85% (i.e. patients with obstructive CAD at ICA [80% of total] + 25% of 20% of patient with non-obstructive CAD [5% of total]).

To accurately estimate this proportion of appropriate ICA the investigators aim to include a sample large enough so that the total width of the 95% confidence interval does not exceed 15%, and thus the maximum margin of error (i.e., the half-width of the confidence interval) does not exceed 7.5%. Assuming a proportion of 85%, the investigators need to include at least 87 patients.

4 TREATMENT OF SUBJECTS Patients will be treated according to current international guidelines and local practice. CMR will be performed as soon as possible prior to ICA (taking into account the requirement of ICA <72 hours after admission) and does not interfere with routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset (>1 hour) chest pain (or angina pectoris equivalent) suspected of non-ST-elevation myocardial infarction (NSTEMI)
* Hospital admission and scheduling for ICA
* Hs-cTn levels meeting the 'observe' criteria (figure 2, p17)
* Age between 18 years - 85 years old
* Written informed consent

Exclusion Criteria:

* Refractory angina or on-going severe ischemia requiring immediate ICA
* Patients requiring ICA < 24 hours after admission (see previous bullet)
* Hemodynamic instability and/or cardiogenic shock (mean arterial pressure <60 mmHg)
* Heart failure (Killip Class ≥ III) requiring intravenously medication (nitroglycerine, diuretics, etc.)
* ST-Elevation Myocardial Infarction (ST-elevation in 2 contiguous leads: ≥0.2mV in men or ≥0.15 mV in women in leads V2-V3 and/or ≥0.1 mV in other leads or new left bundle branch block)
* Symptoms highly suggestive of non-cardiac origin at presentation (as judged by the cardiac ED physician/cardiologist)
* Symptoms highly suggestive of AAD, PE, or acute peri-myocarditis
* Inability to organize ICA and CMR <72 hours after admission (especially for patients admitted on Friday evenings/nights (logistic restrictions).
* Life threatening arrhythmias prior to or during presentation (sustained ventricular tachycardia, repetitive non-sustained ventricular tachycardia, ventricular fibrillation, sinoatrial or atrio-ventricular block)
* Atrial fibrillation with persistent ventricular rate ≥100 beats per minute (bpm) after treatment
* Ongoing tachycardia (≥100/bpm)
* Angina pectoris secondary to anemia (<5.6 mmol/L), untreated hyperthyroidism, or severe hypertension (>200/110 mmHg)
* More than mild aortic and mitral valve calcification or stenosis by latest echocardiography
* Recent revascularization or ACUTE MI (<6 months)
* Known CAD not suitable for further interventions (PCI or CABG)
* Pregnancy
* Breast feeding women
* Life expectancy <1 year (malignancy, etc.)
* Refusal of data storage until 15 years after end of study
* Participation in another investigational study that has not reached its primary endpoint
* Contraindications to CMR:

ODIN-protocol: "Uitvoering van MRI-onderzoek bij patiënten met een cardiaal implanteerbaar elektronisch device (CIED), waaronder een pacemaker en ICD"; ODIN-protocol: "Voorbereiding klinische patiënten voor MRI-onderzoek"

* Metallic implant (vascular clip, neuro-stimulator, cochlear implant)
* Pacemaker or implantable cardiac defibrillator (ICD)
* Claustrophobia
* Body weight >130 kg or body habitus that does not fit into the gantry
* Renal failure (estimated Glomerular Filtration Rate (eGFR) ≤30 mL/min/1,73m2) / chronic renal failure stage 4-5
* Known severe allergy to gadolinium contrast agents (patient with mild allergy is eligible for inclusion when pre-medication according to hospital guidelines can be administered)

  • Contraindications to adenosine:
* High degree atrio-ventricular block (2nd or 3rd degree)
* Severe bronchial asthma
* Chronic obstructive pulmonary disease GOLD >=III
* Concomitant use of Dipyridamole (Persantin®)
* Long QT syndrome (congenital)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the cardiac ED with acute chest pain, a non-diagnostic ERCG, elevated hs-cTn levels meeting the 'observe' criteria, and who are admitted and scheduled for an ICA, will be eligible to participate in this study.
Sampling Method: Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of coronary artery disease as well as non-coronary artery disease related and extra-cardiac diseases | Throuhgout study completion, an expected average of one year
  The prevalence of coronary artery disease as well as non-coronary artery disease related and extra-cardiac diseases in patients presenting with acute chest pain, a non-diagnostic ECG and elevated hs-cTn levels meeting the 'observe' criteria by using CMR early in the diagnostic pathway and at least prior to intended invasive coronary angiography

SECONDARY OUTCOMES:
MACE | 30 days and one year after inclusion
  The number of MACE after 30 days and one year
Composite of MACE and major (non-cardiac) adverse events | 30 days and one year after inclusion
  The number of a composite of MACE and major (non-cardiac) adverse events after 30 days and one year.
Diagnostic accuracy of CMR for the diagnosis of obstructive CAD. | One year after inclusion
  The diagnostic accuracy of CMR for the diagnosis of obstructive CAD (i.e. stenosis ≥70%) by means of specificity and sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhuiya FA, Pitts SR, McCaig LF. Emergency department visits for chest pain and abdominal pain: United States, 1999-2008. NCHS Data Brief. 2010 Sep;(43):1-8. PMID 20854746
- [Background] Fruergaard P, Launbjerg J, Hesse B, Jorgensen F, Petri A, Eiken P, Aggestrup S, Elsborg L, Mellemgaard K. The diagnoses of patients admitted with acute chest pain but without myocardial infarction. Eur Heart J. 1996 Jul;17(7):1028-34. doi: 10.1093/oxfordjournals.eurheartj.a014998. PMID 8809520
- [Background] Lee TH, Goldman L. Evaluation of the patient with acute chest pain. N Engl J Med. 2000 Apr 20;342(16):1187-95. doi: 10.1056/NEJM200004203421607. No abstract available. PMID 10770985
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Pope JH, Ruthazer R, Beshansky JR, Griffith JL, Selker HP. Clinical Features of Emergency Department Patients Presenting with Symptoms Suggestive of Acute Cardiac Ischemia: A Multicenter Study. J Thromb Thrombolysis. 1998 Jul;6(1):63-74. doi: 10.1023/A:1008876322599. PMID 10751787
- [Background] Keller T, Zeller T, Peetz D, Tzikas S, Roth A, Czyz E, Bickel C, Baldus S, Warnholtz A, Frohlich M, Sinning CR, Eleftheriadis MS, Wild PS, Schnabel RB, Lubos E, Jachmann N, Genth-Zotz S, Post F, Nicaud V, Tiret L, Lackner KJ, Munzel TF, Blankenberg S. Sensitive troponin I assay in early diagnosis of acute myocardial infarction. N Engl J Med. 2009 Aug 27;361(9):868-77. doi: 10.1056/NEJMoa0903515. PMID 19710485
- [Background] Reichlin T, Hochholzer W, Bassetti S, Steuer S, Stelzig C, Hartwiger S, Biedert S, Schaub N, Buerge C, Potocki M, Noveanu M, Breidthardt T, Twerenbold R, Winkler K, Bingisser R, Mueller C. Early diagnosis of myocardial infarction with sensitive cardiac troponin assays. N Engl J Med. 2009 Aug 27;361(9):858-67. doi: 10.1056/NEJMoa0900428. PMID 19710484
- [Background] Reichlin T, Twerenbold R, Wildi K, Gimenez MR, Bergsma N, Haaf P, Druey S, Puelacher C, Moehring B, Freese M, Stelzig C, Krivoshei L, Hillinger P, Jager C, Herrmann T, Kreutzinger P, Radosavac M, Weidmann ZM, Pershyna K, Honegger U, Wagener M, Vuillomenet T, Campodarve I, Bingisser R, Miro O, Rentsch K, Bassetti S, Osswald S, Mueller C. Prospective validation of a 1-hour algorithm to rule-out and rule-in acute myocardial infarction using a high-sensitivity cardiac troponin T assay. CMAJ. 2015 May 19;187(8):E243-E252. doi: 10.1503/cmaj.141349. Epub 2015 Apr 13. PMID 25869867
- [Background] Mueller C, Giannitsis E, Christ M, Ordonez-Llanos J, deFilippi C, McCord J, Body R, Panteghini M, Jernberg T, Plebani M, Verschuren F, French J, Christenson R, Weiser S, Bendig G, Dilba P, Lindahl B; TRAPID-AMI Investigators. Multicenter Evaluation of a 0-Hour/1-Hour Algorithm in the Diagnosis of Myocardial Infarction With High-Sensitivity Cardiac Troponin T. Ann Emerg Med. 2016 Jul;68(1):76-87.e4. doi: 10.1016/j.annemergmed.2015.11.013. Epub 2016 Jan 12. PMID 26794254
- [Background] Rubini Gimenez M, Twerenbold R, Jaeger C, Schindler C, Puelacher C, Wildi K, Reichlin T, Haaf P, Merk S, Honegger U, Wagener M, Druey S, Schumacher C, Krivoshei L, Hillinger P, Herrmann T, Campodarve I, Rentsch K, Bassetti S, Osswald S, Mueller C. One-hour rule-in and rule-out of acute myocardial infarction using high-sensitivity cardiac troponin I. Am J Med. 2015 Aug;128(8):861-870.e4. doi: 10.1016/j.amjmed.2015.01.046. Epub 2015 Mar 31. PMID 25840034
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ. 2014 AHA/ACC Guideline for the Management of Patients with Non-ST-Elevation Acute Coronary Syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Dec 23;64(24):e139-e228. doi: 10.1016/j.jacc.2014.09.017. Epub 2014 Sep 23. No abstract available. PMID 25260718
- [Background] Kim HW, Farzaneh-Far A, Kim RJ. Cardiovascular magnetic resonance in patients with myocardial infarction: current and emerging applications. J Am Coll Cardiol. 2009 Dec 29;55(1):1-16. doi: 10.1016/j.jacc.2009.06.059. PMID 20117357
- [Background] Melki D, Lugnegard J, Alfredsson J, Lind S, Eggers KM, Lindahl B, Jernberg T. Implications of Introducing High-Sensitivity Cardiac Troponin T Into Clinical Practice: Data From the SWEDEHEART Registry. J Am Coll Cardiol. 2015 Apr 28;65(16):1655-1664. doi: 10.1016/j.jacc.2015.02.044. PMID 25908071
- [Background] Plein S, Greenwood JP, Ridgway JP, Cranny G, Ball SG, Sivananthan MU. Assessment of non-ST-segment elevation acute coronary syndromes with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Dec 7;44(11):2173-81. doi: 10.1016/j.jacc.2004.08.056. PMID 15582315
- [Background] Cury RC, Shash K, Nagurney JT, Rosito G, Shapiro MD, Nomura CH, Abbara S, Bamberg F, Ferencik M, Schmidt EJ, Brown DF, Hoffmann U, Brady TJ. Cardiac magnetic resonance with T2-weighted imaging improves detection of patients with acute coronary syndrome in the emergency department. Circulation. 2008 Aug 19;118(8):837-44. doi: 10.1161/CIRCULATIONAHA.107.740597. Epub 2008 Aug 4. PMID 18678772
- [Background] Danad I, Szymonifka J, Twisk JWR, Norgaard BL, Zarins CK, Knaapen P, Min JK. Diagnostic performance of cardiac imaging methods to diagnose ischaemia-causing coronary artery disease when directly compared with fractional flow reserve as a reference standard: a meta-analysis. Eur Heart J. 2017 Apr 1;38(13):991-998. doi: 10.1093/eurheartj/ehw095. PMID 27141095
- [Background] Greenwood JP, Ripley DP, Berry C, McCann GP, Plein S, Bucciarelli-Ducci C, Dall'Armellina E, Prasad A, Bijsterveld P, Foley JR, Mangion K, Sculpher M, Walker S, Everett CC, Cairns DA, Sharples LD, Brown JM; CE-MARC 2 Investigators. Effect of Care Guided by Cardiovascular Magnetic Resonance, Myocardial Perfusion Scintigraphy, or NICE Guidelines on Subsequent Unnecessary Angiography Rates: The CE-MARC 2 Randomized Clinical Trial. JAMA. 2016 Sep 13;316(10):1051-60. doi: 10.1001/jama.2016.12680. PMID 27570866
- [Background] Kim RJ, Farzaneh-Far A. The diagnostic utility of cardiovascular magnetic resonance in patients with chest pain, elevated cardiac enzymes and non-obstructed coronary arteries. Rev Esp Cardiol. 2009 Sep;62(9):966-71. doi: 10.1016/s1885-5857(09)73261-x. No abstract available. English, Spanish. PMID 19712616
- [Background] Assomull RG, Lyne JC, Keenan N, Gulati A, Bunce NH, Davies SW, Pennell DJ, Prasad SK. The role of cardiovascular magnetic resonance in patients presenting with chest pain, raised troponin, and unobstructed coronary arteries. Eur Heart J. 2007 May;28(10):1242-9. doi: 10.1093/eurheartj/ehm113. Epub 2007 May 3. PMID 17478458
- [Background] Pathik B, Raman B, Mohd Amin NH, Mahadavan D, Rajendran S, McGavigan AD, Grover S, Smith E, Mazhar J, Bridgman C, Ganesan AN, Selvanayagam JB. Troponin-positive chest pain with unobstructed coronary arteries: incremental diagnostic value of cardiovascular magnetic resonance imaging. Eur Heart J Cardiovasc Imaging. 2016 Oct;17(10):1146-52. doi: 10.1093/ehjci/jev289. Epub 2015 Nov 20. PMID 26590396
- [Background] Revel MP, Sanchez O, Couchon S, Planquette B, Hernigou A, Niarra R, Meyer G, Chatellier G. Diagnostic accuracy of magnetic resonance imaging for an acute pulmonary embolism: results of the 'IRM-EP' study. J Thromb Haemost. 2012 May;10(5):743-50. doi: 10.1111/j.1538-7836.2012.04652.x. PMID 22321816
- [Background] Smulders MW, Kietselaer BL, Das M, Wildberger JE, Crijns HJ, Veenstra LF, Brunner-La Rocca HP, van Dieijen-Visser MP, Mingels AM, Dagnelie PC, Post MJ, Gorgels AP, van Asselt AD, Vogel G, Schalla S, Kim RJ, Bekkers SC. The role of cardiovascular magnetic resonance imaging and computed tomography angiography in suspected non-ST-elevation myocardial infarction patients: design and rationale of the CARdiovascular Magnetic rEsoNance imaging and computed Tomography Angiography (CARMENTA) trial. Am Heart J. 2013 Dec;166(6):968-75. doi: 10.1016/j.ahj.2013.09.012. Epub 2013 Oct 23. PMID 24268210
- [Background] Bruder O, Schneider S, Nothnagel D, Pilz G, Lombardi M, Sinha A, Wagner A, Dill T, Frank H, van Rossum A, Schwitter J, Nagel E, Senges J, Sabin G, Sechtem U, Mahrholdt H. Acute adverse reactions to gadolinium-based contrast agents in CMR: multicenter experience with 17,767 patients from the EuroCMR Registry. JACC Cardiovasc Imaging. 2011 Nov;4(11):1171-6. doi: 10.1016/j.jcmg.2011.06.019. PMID 22093267
- [Background] Bruder O, Wagner A, Lombardi M, Schwitter J, van Rossum A, Pilz G, Nothnagel D, Steen H, Petersen S, Nagel E, Prasad S, Schumm J, Greulich S, Cagnolo A, Monney P, Deluigi CC, Dill T, Frank H, Sabin G, Schneider S, Mahrholdt H. European Cardiovascular Magnetic Resonance (EuroCMR) registry--multi national results from 57 centers in 15 countries. J Cardiovasc Magn Reson. 2013 Jan 18;15(1):9. doi: 10.1186/1532-429X-15-9. PMID 23331632
- [Background] Burg MA, Lopez ED, Dailey A, Keller ME, Prendergast B. The potential of survivorship care plans in primary care follow-up of minority breast cancer patients. J Gen Intern Med. 2009 Nov;24 Suppl 2(Suppl 2):S467-71. doi: 10.1007/s11606-009-1012-y. PMID 19838852
- [Background] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Circulation. 2002 Jan 29;105(4):539-42. doi: 10.1161/hc0402.102975. No abstract available. PMID 11815441
- [Background] Forsting M, Palkowitsch P. Prevalence of acute adverse reactions to gadobutrol--a highly concentrated macrocyclic gadolinium chelate: review of 14,299 patients from observational trials. Eur J Radiol. 2010 Jun;74(3):e186-92. doi: 10.1016/j.ejrad.2009.06.005. Epub 2009 Jul 2. PMID 19574008
- [Background] Ingkanisorn WP, Kwong RY, Bohme NS, Geller NL, Rhoads KL, Dyke CK, Paterson DI, Syed MA, Aletras AH, Arai AE. Prognosis of negative adenosine stress magnetic resonance in patients presenting to an emergency department with chest pain. J Am Coll Cardiol. 2006 Apr 4;47(7):1427-32. doi: 10.1016/j.jacc.2005.11.059. Epub 2006 Mar 20. PMID 16580532
- [Background] Cerqueira MD, Verani MS, Schwaiger M, Heo J, Iskandrian AS. Safety profile of adenosine stress perfusion imaging: results from the Adenoscan Multicenter Trial Registry. J Am Coll Cardiol. 1994 Feb;23(2):384-9. doi: 10.1016/0735-1097(94)90424-3. PMID 8294691
- [Background] Wahl A, Paetsch I, Gollesch A, Roethemeyer S, Foell D, Gebker R, Langreck H, Klein C, Fleck E, Nagel E. Safety and feasibility of high-dose dobutamine-atropine stress cardiovascular magnetic resonance for diagnosis of myocardial ischaemia: experience in 1000 consecutive cases. Eur Heart J. 2004 Jul;25(14):1230-6. doi: 10.1016/j.ehj.2003.11.018. PMID 15246641